CLINICAL TRIAL: NCT03780101
Title: Pathology and Imaging in Kidney Allografts
Acronym: PIKA
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulties due to impact of COVID-19 pandemic
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN18RE474; 248675 (Other: IRAS project ID)
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Renal Transplant Rejection; Chronic Kidney Diseases; Fibrosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fibrosis biomarkers, which may include galactin-3, microRNA (including miR-214, miR-21 and miR-29), tissue inhibitor metalloproteinases (TIMP)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multi-parametric renal MRI — Multi-parametric functional magnetic resonance imaging of a transplant kidney including sequences for T1, T2, diffusion-weighted imaging, diffusion tensor imaging and arterial spin labelling.

SUMMARY:
This study will perform multi-parametric renal MRI in 70 patients with a renal transplant who are undergoing a clinically indicated biopsy of their transplant. The aim of this study is to compare findings on renal MRI with those seen on histology.

DETAILED DESCRIPTION:
Background: Renal transplantation is the optimal treatment for patients with renal failure. However, transplant life-span is finite and commonly limited due to the development of chronic rejection and other causes of irreversible fibrosis. At present, renal transplant biopsy is required to diagnose the cause of transplant dysfunction. Renal biopsies are invasive procedures that carry risks of bleeding, damage to the transplant and discomfort to patients. Functional magnetic resonance imaging (MRI) of the kidneys is an emerging field of research that has potential to non-invasively define and quantify parenchymal renal disease including fibrosis and inflammation. There is a paucity of data correlating multi-parametric renal MRI sequences with histological findings on biopsy, especially in patients with renal transplants.

Study participants: 70 adult renal transplant recipients who have been referred for a clinically indicated biopsy of their transplant kidney.

Study design: Participants will undergo multi-parametric renal MRI at time of biopsy. In patients who receive treatment for acute rejection, a second renal MRI will be undertaken at completion of treatment. Blood tests for fibrosis biomarkers and routine clinical measures of transplant function will be obtained at time of MRI scanning.

Objectives:

1. Assess the correlation between functional renal MRI sequences and histological markers of fibrosis and inflammation.
2. Assess the change in functional MRI sequences in response to treatment for acute rejection in renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Recipient of a kidney transplant
* Referred for clinically indicated biopsy of transplant kidney
* Ability to comply with study procedures.
* Ability to give informed consent.

Exclusion Criteria:

* Any contraindication to MRI
* Known pregnancy or intent to conceive during the study period
* Clinical suspicion of delayed graft function as the cause of transplant dysfunction
* Any other reason considered by a study physician to make the subject inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant recipients referred for a clinically-indicated biopsy of their transplant kidney
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Comparison of MRI biomarkers for fibrosis with histology | Baseline
  Correlation between diffusion weighted imaging on renal MRI and reported percentage of cortical area on biopsy showing interstitial fibrosis.

SECONDARY OUTCOMES:
Renal MRI following treatment for acute rejection | 2 weeks
  Correlation between change in native T1 and serum creatinine following treatment for acute rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Alastair J Rankin, MBChB, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow & Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided